CLINICAL TRIAL: NCT02178306
Title: An Open-labeled, Placebo run-in, Multicentre Study to Investigate the Efficacy and Safety of Telmisartan (40 and 80 mg QD p.o.) in 3 Strata of Mild to Moderate Hypertensive Patients (Sitting Diastolic Blood Pressure ≥ 90 mmHg and ≤ 109 mmHg From Office Cuff Measurement) With Mild/Moderate or Severe Renal Impairment or Requiring Maintenance Hemodialysis. (ESPRIT Study = Efficacy and Safety in Patients With Renal Impairment Treated With Telmisartan)
Brief Title: Efficacy and Safety of Telmisartan in Hypertensive Patients With Mild/Moderate or Severe Renal Impairment or Requiring Hemodialysis
Acronym: ESPRIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 502.339
Record Dates: First submitted 2014-06-27; First posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

ARMS (1):
- Telmisartan (Experimental)
  Interventions: Drug: Telmisartan low dose; Drug: Telmisartan high dose; Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan low dose
Drug: Telmisartan high dose — patients switch to high dose if mean SBP >= 85 mmHg after 4 weeks of treatment
Drug: Placebo — Run-in phase

SUMMARY:
To evaluate the safety and efficacy, in particular with regard to renal function of telmisartan at the doses of 40 mg and 80 mg in hypertensive patients with moderate to endstage renal impairment after 12 weeks of treatment

ELIGIBILITY:
Inclusion Criteria:

1. Mild to moderate hypertension, sitting diastolic BP ≥ 90 mmHg and BP ≤ 109 mmHg at visit 2
2. No increase of serum creatinine over 30% within 6 months before the trial
3. Stable renal insufficiency with a serum creatinine between 200 and 600 µmol/l or maintenance of hemodialysis
4. Stable proteinuria of at least 500 mg/24h
5. No change in hemodialysis regimen within the last two months prior to visit 1
6. 18 years of age or more
7. Ability to provide written informed consent in accordance with good clinical practice and local registration
8. Able to stop current antihypertensive therapy (ACE-Inhibitors or angiotensin II receptor subtype 1- Blocker) without risk to the patient

Exclusion Criteria:

1. Pre-menopausal women (last menstruation ≤ 1 year prior to start of run-in-phase) who:

   1. are not surgically sterile; and/or
   2. are nursing
   3. are of child-bearing potential and are NOT practicing acceptable means of birth control, do NOT plan to continue using this method throughout the study and do NOT agree to submit to periodic pregnancy testing during participation in studies of ≥ 3-months duration. Acceptable methods of birth control include oral, implantable or injectable contraceptives
2. Known or suspected renovascular hypertension
3. Mean sitting SBP ≥ 180 mmHg or mean sitting DBP ≥110 mmHg during any visit of the placebo run-in phase
4. Hepatic dysfunction as defined by the following laboratory parameters:

   serum glutamate pyruvate transaminase (ALT) or serum glutamate oxaloacetate transaminase (AST) > than 2 times the upper limit of normal range
5. Bilateral renal artery stenosis; renal artery stenosis in a solitary kidney, patients postrenal transplant or with only one kidney
6. Clinically relevant hypo- or hyperkalaemia
7. Uncorrected volume depletion
8. Uncorrected sodium depletion
9. Primary aldosteronism
10. Hereditary fructose intolerance
11. Biliary obstructive disorders
12. Patients who have previously experienced symptoms characteristic of angioedema during treatment with ACE inhibitors or angiotensin II antagonists
13. History of drug or alcohol abuse within 6 months
14. Chronic administration of any medications known to affect blood pressure, except medication allowed by the protocol (ß-blocker, alpha-blocker, calcium antagonists, clonidine, minoxidil, and diuretics)
15. Any investigational therapy within one month of signing the informed consent form
16. Known hypersensitivity to any component of the formulation
17. Has no contra-indication to a placebo run-in period (e.g. unstable angina within the past 3 months, stroke within the past 6 months or myocardial infarction or cardiac surgery within the past 3 months)
18. Any other clinical condition which, in the opinion of the investigator, would not allow safe completion of the protocol and safe administration of telmisartan
19. Compliance < 70% during run-in period (defined by pill count)
20. History of heart failure, malignancy, or any disorders requiring immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2000-09; Primary Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in seated diastolic blood pressure (DBP) at trough | 12 weeks after start of treatment

SECONDARY OUTCOMES:
Change from baseline in seated systolic blood pressure (SBP) at trough | 12 weeks after start of treatment
Frequency of response categories of blood pressure | After 12 weeks of treatment
  Categories:
  1. BP normal
  2. DBP control
  3. DBP response
  4. SBP response
  5. BP high normal
Changes from baseline in proteinuria | 12 weeks after start of treatment
Change in electrolyte excretion | 12 weeks after start of treatment
Area under the telmisartan plasma concentration-time curve | Day 7 and 12 weeks after start of treatment
Maximum plasma concentration (Cmax) of telmisartan | Day 7 and 12 weeks after start of treatment
Time to peak (Tmax) plasma concentrations of telmisartan | Day 7 and 12 weeks after start of treatment
Extent of protein binding of telmisartan | Day 7 and 12 weeks after start of treatment
  equilibrium dialysis with subsequent determination of protein-bound telmisartan fraction